CLINICAL TRIAL: NCT02527278
Title: A Retrospective Claims Analysis to Calculate the Proportion of Women Undergoing Hysterectomy, Salpingectomy, Salpingostomy, Hysteroscopy or Who Had a Diagnosis of Pelvic Pain After Hysteroscopic Sterilization or Laparoscopic Tubal Ligation
Brief Title: Retrospective Claims Analysis of Hysterectomy After Sterilization
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18477
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Laparoscopic tubal ligation (no pain): Women who have laparoscopic tubal ligation, with no previous diagnosis of pain at baseline
  Interventions: Procedure: Laparoscopic tubal ligation
- Laparoscopic tubal ligation (pain): Women who have laparoscopic tubal ligation, with a previous diagnosis of pain at baseline
  Interventions: Procedure: Laparoscopic tubal ligation
- Hysteroscopic sterilization (no pain): Women who have hysteroscopic sterilization, with no previous diagnosis of pain at baseline
  Interventions: Procedure: Hysteroscopic sterilization
- Hysteroscopic sterilization (pain): Women who have hysteroscopic sterilization, with a previous diagnosis of pain at baseline
  Interventions: Procedure: Hysteroscopic sterilization

INTERVENTIONS:
Procedure: Laparoscopic tubal ligation — Female permanent birth control method performed via a surgical procedure
  Groups: Laparoscopic tubal ligation (no pain); Laparoscopic tubal ligation (pain)
Procedure: Hysteroscopic sterilization — Female permanent birth control method performed via placement of a device
  Groups: Hysteroscopic sterilization (no pain); Hysteroscopic sterilization (pain)

SUMMARY:
The research questions are:

1. What is the proportion of women undergoing hysterectomy after hysteroscopic sterilization or laparoscopic tubal ligation?
2. What is the proportion of women undergoing salpingectomy, salpingostomy, or hysteroscopy after hysteroscopic sterilization or laparoscopic tubal ligation?
3. What is the proportion of women who have a diagnosis of pelvic pain after hysteroscopic sterilization or laparoscopic tubal ligation?

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 through 49 years at the index date
* at least one claim of the hysteroscopic sterilization procedure or interval laparoscopic tubal ligation at any time during January 1, 2010 -December 31, 2012
* Had 6 months of continuous medical and pharmacy benefits pre-index date which is considered the baseline period to capture all patient characteristics prior to the procedure
* Had 12 months of continuous medical and pharmacy benefits post-index date (i.e., follow-up period)

Exclusion Criteria:

* Women who underwent a postpartum tubal ligation procedure during the entire study period
* Women who had claims of a sterilization procedure during the baseline period
* Women who had a claim for pregnancy or delivery within 6 weeks prior to the index date
* Women who had more than one type of sterilization procedure (i.e., combination of hysteroscopic sterilization, laparoscopic tubal ligation or mini-laparotomy) on the same index date
* Women who had concurrent procedures on the same day as the index sterilization procedure that were performed for reasons beyond the purpose of sterilization

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 18 - 49 at the time of the sterilization procedure from an administrative claims database
Sampling Method: Non-Probability Sample
Enrollment: 19317 (Actual)
Dates: Start 2015-07-30 (Actual); Primary Completion 2016-02-09 (Actual); Study Completion 2016-02-09 (Actual)

PRIMARY OUTCOMES:
Proportion of women undergoing hysterectomy after hysteroscopic sterilization or laparoscopic tubal ligation | Within 12 months after the procedure

SECONDARY OUTCOMES:
Proportion of women undergoing salpingectomy after hysteroscopic sterilization or laparoscopic tubal ligation | Within 12 months after the procedure
Proportion of women undergoing salpingostomy after hysteroscopic sterilization or laparoscopic tubal ligation | Within 12 months after the procedure
Proportion of women undergoing hysteroscopy after hysteroscopic sterilization or laparoscopic tubal ligation | Within 12 months after the procedure
Proportion of women who have a diagnosis of pelvic pain after hysteroscopic sterilization or laparoscopic tubal ligation | Within 12 months after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Whippany, New Jersey, United States